CLINICAL TRIAL: NCT05296213
Title: Medical Treatment of Early-Enamel Carious Lesion Using Different Remeneralizing Agents: 2-years Randomized Clinical Trial
Brief Title: Medical Treatment of Early-Enamel Carious Lesion Using Different Remeneralizing Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M03060819
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Enamel Caries
Keywords: Enamel remineralization; Randomized Clinical Trial; Experimental Tricalcium silicate; Sillver diamine flouride-potassium iodide
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- silver diamine fluoride-potassium iodide SDF-KI (riva star) (Experimental): SDF-KI was applied once as a professional application over the early enamel lesions in cervical third of the buccal surface of molar teeth.
  Interventions: Drug: Silver diamine fluoride- potassium iodide
- casein phosphopeptide amorphous calcium phosphate CPP-ACP(tooth mousse) (Experimental): CPP-ACP cream was applied twice daily according to manufacturer's instructions over the early enamel lesions in cervical third of the buccal surface of molar teeth.
  Interventions: Drug: Casein phosphopeptide amorphous calcium phosphate
- Experimental tricalcium silicate (Experimental): Experimental tricalcium silicate paste was applied twice daily over the early enamel lesions in cervical third of the buccal surface of molar teeth
  Interventions: Drug: experimental tricalcium silicate

INTERVENTIONS:
Drug: Silver diamine fluoride- potassium iodide — SDF-KI (riva star, SDI.Ltd )was applied ( as a professional application) by micro brush over the early enamel lesions on the buccal surface of molar teeth
  Arms: silver diamine fluoride-potassium iodide SDF-KI (riva star)
Drug: Casein phosphopeptide amorphous calcium phosphate — CPP-ACP (tooth mousse, GC, Matraville Sydney, Australia) was applied by using micro brush over the early enamel lesions on the buccal surface of the molar teeth twice daily. the patients were instructed to leave it for about 3minutes before rinsing
  Arms: casein phosphopeptide amorphous calcium phosphate CPP-ACP(tooth mousse)
Drug: experimental tricalcium silicate — prepared tricalcium silicate paste was applied by using micro brush over the early enamel lesions on the buccal surface of the molar teeth twice daily. the patients were instructed to leave it for about 3minutes before rinsing
  Arms: Experimental tricalcium silicate

SUMMARY:
Medical Treatment of Early-Enamel Carious Lesion using Different Remeneralizing agents

DETAILED DESCRIPTION:
Medical management of incipient lesions by application of remineralizing agents like fluoride therapy, amorphous calcium phosphate (ACP), and Casin phosphopeptide amorphous calcium phosphate (CPP-ACP) has proved to be effective in reversing such lesions.

Fluoride was considered the "gold standard" remineralizing agent , However several recent researchers found that; the ideal remineralizing agents should diffuse or deliver calcium and phosphate ions into early enamel lesion.

Calcium-silicate based material such as β-CaSiO3 and β-Ca2SiO4 play an important role in hard tissue regeneration, showing good bioactivity and biocompatibility and can induce bone like apetite formation in stimulated body fluids. when β-CaSiO3 and β-Ca2SiO4 come in contact with saliva it will be dissolve forming silanol group (Si-O ) on the enamel surface which can bind to Ca ions and inducing the precipitation of hydroxyapatite.

In the light of this, this study was designed to compare the remineralization potential of silver diamine flouride/ potassium iodide, casin phosphopeptide amorphous calcium phosphate and experimental tricalcium silicate on early enamel lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early enamel lesions (ICDAS score 1 and 2).
* Patients with normal occlusion .
* Patients must have a good oral hygiene
* patients free from any systemic diseases and don't receive any medication

Exclusion Criteria:

* smoker patients
* pregnant females
* patients with bad oral hygiene
* patients with enamel defects ( Amelogenesis Imperfecta, fluorosis, cracks or any developmental defects)

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Medical Treatment of Early-Enamel Carious Lesion using Different Remeneralizing agents | 2-years after the first application of the remineralizing agents
  The primary outcome was the change in laser fluorescence values that was detected by DIAGNODent Pen. The obtained values were interpreted according to the scale provided by the manufacture:
  * Value between (0-13) refers to sound enamel substrate
  * Value between (14-20) refers to early enamel caries

CONTACTS AND LOCATIONS:
Locations (1):
- Kareem Hamdi, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 3 Months for 5 years
Access Criteria: for every one